CLINICAL TRIAL: NCT04793828
Title: The Effect of a Transdiagnostic, Self-guided Internet Intervention ("Velibra") for Waitlist Patients With Anxiety Disorders
Brief Title: A Transdiagnostic, Self-guided Internet Intervention ("Velibra") for Waitlist Patients With Anxiety Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Lena Pyrkosch, Psychologist, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA 1/322/19
Record Dates: First submitted 2021-02-22; First posted 2021-03-11 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Panic Disorder With Agoraphobia; Panic Disorder Without Agoraphobia; Generalized Anxiety Disorder; Social Anxiety Disorder
Keywords: cognitive behavioral therapy; internet intervention; administrative-supported; anxiety; panic disorder; social anxiety disorder; generalized anxiety disorder; computerized CBT; anxiety disorders; velibra; psychotherapy
MeSH Terms: conditions — Generalized Anxiety Disorder; Phobia, Social; Anxiety Disorders; Panic Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (velibra) (Experimental): Arm consisting of participants who receive velibra, an internet-based cognitive behavioral therapy program.
  Interventions: Behavioral: Velibra

INTERVENTIONS:
Behavioral: Velibra — Velibra is an internet-based cognitive behavioral therapy program developed by GAIA AG. It consists of six modules which are meant to be completed over a span of 6 weeks. The first module educates participants about anxiety and the treatment program. The second module focuses on cognitive techniques for dealing with anxiety. In the third module, relaxation techniques are practiced. The fourth module encourages the participant to practice non-anxious behaviors. In the fifth module, the central topic is the experience of social situations in non-anxious ways. The sixth and final module consists of a summary and recapitulation of the most important content.

SUMMARY:
The project's aim is to investigate the effect of a transdiagnostic, self-guided, internet-based cognitive behavioral therapy program in waitlist patients with anxiety disorders.

DETAILED DESCRIPTION:
Patients who fulfill the inclusion criteria and are interested in psychotherapy are offered participation in the study to bridge the waiting time for face-to-face psychotherapy. After obtaining informed consent, a pre-treatment assessment is conducted. Then, participants are provided access to velibra, an internet-based cognitive behavioral therapy program which they can work through at their own pace. While velibra is a self-guided program, participants are supported by study personnel during four assessments at four time points: pre-treatment, mid-treatment (after the first three velibra modules), post-treatment and at the one-month follow-up. The investigators expect improvements on the primary as well as the secondary outcomes. Furthermore, the investigators are interested in studying the acceptability of velibra and whether positive changes already become observable after the first three modules, i.e., at the mid-treatment assessment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of panic disorder with or without agoraphobia, social anxiety disorder, or generalized anxiety disorder
* Knowledge of German that is sufficient for engaging with the treatment and responding to the questionnaires
* Written informed consent
* Internet access

Exclusion Criteria:

* Diagnoses of severe mental comorbidities (e.g., schizophrenia, severe major depression, borderline personality disorder)
* Acute suicidality
* Started or changed anxiolytic pharmacotherapy recently (currently or in the past four weeks)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Panic and Agoraphobia Scale (PAS) | Baseline (pre-treatment)
  The Panic and Agoraphobia Scale (PAS) is a self-report questionnaire used to measure the symptom severity of panic disorder with or without agoraphobia. It is given to study participants diagnosed with panic disorder with or without agoraphobia. Total score values range from 0 to 52, with higher scores indicating a worse outcome.
Panic and Agoraphobia Scale (PAS) | During the intervention (mid-treatment)
  The Panic and Agoraphobia Scale (PAS) is a self-report questionnaire used to measure the symptom severity of panic disorder with or without agoraphobia. It is given to study participants diagnosed with panic disorder with or without agoraphobia. Total score values range from 0 to 52, with higher scores indicating a worse outcome.
Panic and Agoraphobia Scale (PAS) | Immediately after / as soon as possible after the intervention (post-treatment)
  The Panic and Agoraphobia Scale (PAS) is a self-report questionnaire used to measure the symptom severity of panic disorder with or without agoraphobia. It is given to study participants diagnosed with panic disorder with or without agoraphobia. Total score values range from 0 to 52, with higher scores indicating a worse outcome.
Panic and Agoraphobia Scale (PAS) | 1-month follow-up
  The Panic and Agoraphobia Scale (PAS) is a self-report questionnaire used to measure the symptom severity of panic disorder with or without agoraphobia. It is given to study participants diagnosed with panic disorder with or without agoraphobia. Total score values range from 0 to 52, with higher scores indicating a worse outcome.
Liebowitz Social Anxiety Scale (LSAS) | Baseline (pre-treatment)
  The Liebowitz Social Anxiety Scale (LSAS) is a self-report questionnaire used to measure the symptom severity of social anxiety disorder. It is given to study participants diagnosed with social anxiety disorder. Total score values range from 0 to 72, with higher scores indicating a worse outcome.
Liebowitz Social Anxiety Scale (LSAS) | During the intervention (mid-treatment)
  The Liebowitz Social Anxiety Scale (LSAS) is a self-report questionnaire used to measure the symptom severity of social anxiety disorder. It is given to study participants diagnosed with social anxiety disorder. Total score values range from 0 to 72, with higher scores indicating a worse outcome.
Liebowitz Social Anxiety Scale (LSAS) | Immediately after / as soon as possible after the intervention (post-treatment)
  The Liebowitz Social Anxiety Scale (LSAS) is a self-report questionnaire used to measure the symptom severity of social anxiety disorder. It is given to study participants diagnosed with social anxiety disorder. Total score values range from 0 to 72, with higher scores indicating a worse outcome.
Liebowitz Social Anxiety Scale (LSAS) | 1-month follow-up
  The Liebowitz Social Anxiety Scale (LSAS) is a self-report questionnaire used to measure the symptom severity of social anxiety disorder. It is given to study participants diagnosed with social anxiety disorder. Total score values range from 0 to 72, with higher scores indicating a worse outcome.
Penn State Worry Questionnaire (PSWQ) | Baseline (pre-treatment)
  The Penn State Worry Questionnaire (PSWQ) is a self-report questionnaire used to measure the symptom severity of generalized anxiety disorder It is given to study participants diagnosed with generalized anxiety disorder. Total score values range from 16 to 80, with higher scores indicating a worse outcome.
Penn State Worry Questionnaire (PSWQ) | During the intervention (mid-treatment)
  The Penn State Worry Questionnaire (PSWQ) is a self-report questionnaire used to measure the symptom severity of generalized anxiety disorder It is given to study participants diagnosed with generalized anxiety disorder. Total score values range from 16 to 80, with higher scores indicating a worse outcome.
Penn State Worry Questionnaire (PSWQ) | Immediately after / as soon as possible after the intervention (post-treatment)
  The Penn State Worry Questionnaire (PSWQ) is a self-report questionnaire used to measure the symptom severity of generalized anxiety disorder It is given to study participants diagnosed with generalized anxiety disorder. Total score values range from 16 to 80, with higher scores indicating a worse outcome.
Penn State Worry Questionnaire (PSWQ) | 1-month follow-up
  The Penn State Worry Questionnaire (PSWQ) is a self-report questionnaire used to measure the symptom severity of generalized anxiety disorder It is given to study participants diagnosed with generalized anxiety disorder. Total score values range from 16 to 80, with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Baseline (pre-treatment)
  The Beck Anxiety Inventory (BAI) is a self-report questionnaire used to measure the symptom severity of anxiety in general. It is given to all study participants regardless of diagnosis. Total score values range from 0 to 63, with higher scores indicating a worse outcome.
Beck Anxiety Inventory (BAI) | During the intervention (mid-treatment)
  The Beck Anxiety Inventory (BAI) is a self-report questionnaire used to measure the symptom severity of anxiety in general. It is given to all study participants regardless of diagnosis. Total score values range from 0 to 63, with higher scores indicating a worse outcome.
Beck Anxiety Inventory (BAI) | Immediately after / as soon as possible after the intervention (post-treatment)
  The Beck Anxiety Inventory (BAI) is a self-report questionnaire used to measure the symptom severity of anxiety in general. It is given to all study participants regardless of diagnosis. Total score values range from 0 to 63, with higher scores indicating a worse outcome.
Beck Anxiety Inventory (BAI) | 1-month follow-up
  The Beck Anxiety Inventory (BAI) is a self-report questionnaire used to measure the symptom severity of anxiety in general. It is given to all study participants regardless of diagnosis. Total score values range from 0 to 63, with higher scores indicating a worse outcome.
Beck Depression Inventory-II (BDI-II) | Baseline (pre-treatment)
  The Beck Depression Inventory-II (BDI-II) is a self-report questionnaire used to measure the symptom severity of depression. It is given to all study participants regardless of diagnosis. Total score values range from 0 to 63, with higher scores indicating a worse outcome.
Beck Depression Inventory-II (BDI-II) | During the intervention (mid-treatment)
  The Beck Depression Inventory-II (BDI-II) is a self-report questionnaire used to measure the symptom severity of depression. It is given to all study participants regardless of diagnosis. Total score values range from 0 to 63, with higher scores indicating a worse outcome.
Beck Depression Inventory-II (BDI-II) | Immediately after / as soon as possible after the intervention (post-treatment)
  The Beck Depression Inventory-II (BDI-II) is a self-report questionnaire used to measure the symptom severity of depression. It is given to all study participants regardless of diagnosis. Total score values range from 0 to 63, with higher scores indicating a worse outcome.
Beck Depression Inventory-II (BDI-II) | 1-month follow-up
  The Beck Depression Inventory-II (BDI-II) is a self-report questionnaire used to measure the symptom severity of depression. It is given to all study participants regardless of diagnosis. Total score values range from 0 to 63, with higher scores indicating a worse outcome.
Anxiety Sensitivity Index (ASI) | Baseline (pre-treatment)
  The Anxiety Sensitivity Index (ASI) is a self-report questionnaire used to measure anxiety sensitivity. It is given to all study participants regardless of diagnosis. Total score values range from 0 to 64, with higher scores indicating a worse outcome.
Anxiety Sensitivity Index (ASI) | During the intervention (mid-treatment)
  The Anxiety Sensitivity Index (ASI) is a self-report questionnaire used to measure anxiety sensitivity. It is given to all study participants regardless of diagnosis. Total score values range from 0 to 64, with higher scores indicating a worse outcome.
Anxiety Sensitivity Index (ASI) | Immediately after / as soon as possible after the intervention (post-treatment)
  The Anxiety Sensitivity Index (ASI) is a self-report questionnaire used to measure anxiety sensitivity. It is given to all study participants regardless of diagnosis. Total score values range from 0 to 64, with higher scores indicating a worse outcome.
Anxiety Sensitivity Index (ASI) | 1-month follow-up
  The Anxiety Sensitivity Index (ASI) is a self-report questionnaire used to measure anxiety sensitivity. It is given to all study participants regardless of diagnosis. Total score values range from 0 to 64, with higher scores indicating a worse outcome.
ICD-10-Symptom-Rating (ISR) | Baseline (pre-treatment)
  The ICD-10-Symptom-Rating (ISR) is a self-report questionnaire used to measure mental distress related to syndromes defined in the ICD-10. It is given to all study participants regardless of diagnosis. Total score values (based on subscale means) range from 0 to 4, with higher scores indicating a worse outcome.
ICD-10-Symptom-Rating (ISR) | During the intervention (mid-treatment)
  The ICD-10-Symptom-Rating (ISR) is a self-report questionnaire used to measure mental distress related to syndromes defined in the ICD-10. It is given to all study participants regardless of diagnosis. Total score values (based on subscale means) range from 0 to 4, with higher scores indicating a worse outcome.
ICD-10-Symptom-Rating (ISR) | Immediately after / as soon as possible after the intervention (post-treatment)
  The ICD-10-Symptom-Rating (ISR) is a self-report questionnaire used to measure mental distress related to syndromes defined in the ICD-10. It is given to all study participants regardless of diagnosis. Total score values (based on subscale means) range from 0 to 4, with higher scores indicating a worse outcome.
ICD-10-Symptom-Rating (ISR) | 1-month follow-up
  The ICD-10-Symptom-Rating (ISR) is a self-report questionnaire used to measure mental distress related to syndromes defined in the ICD-10. It is given to all study participants regardless of diagnosis. Total score values (based on subscale means) range from 0 to 4, with higher scores indicating a worse outcome.
Short-Form Health Survey (SF-12) | Baseline (pre-treatment)
  The Short-Form Health Survey (SF-12) is a self-report questionnaire used to measure health-related quality of life. It is given to all study participants regardless of diagnosis. Values of the summary scores range from 0 to 100, with higher scores indicating a better outcome.
Short-Form Health Survey (SF-12) | During the intervention (mid-treatment)
  The Short-Form Health Survey (SF-12) is a self-report questionnaire used to measure health-related quality of life. It is given to all study participants regardless of diagnosis. Values of the summary scores range from 0 to 100, with higher scores indicating a better outcome.
Short-Form Health Survey (SF-12) | Immediately after / as soon as possible after the intervention (post-treatment)
  The Short-Form Health Survey (SF-12) is a self-report questionnaire used to measure health-related quality of life. It is given to all study participants regardless of diagnosis. Values of the summary scores range from 0 to 100, with higher scores indicating a better outcome.
Short-Form Health Survey (SF-12) | 1-month follow-up
  The Short-Form Health Survey (SF-12) is a self-report questionnaire used to measure health-related quality of life. It is given to all study participants regardless of diagnosis. Values of the summary scores range from 0 to 100, with higher scores indicating a better outcome.
General Self--Efficacy Scale (GES) | Baseline (pre-treatment)
  The General Self--Efficacy Scale (GES) is a self-report questionnaire used to measure self-efficacy. It is given to all study participants regardless of diagnosis. Total score values range from 10 to 40, with higher scores indicating a better outcome.
General Self--Efficacy Scale (GES) | During the intervention (mid-treatment)
  The General Self--Efficacy Scale (GES) is a self-report questionnaire used to measure self-efficacy. It is given to all study participants regardless of diagnosis. Total score values range from 10 to 40, with higher scores indicating a better outcome.
General Self--Efficacy Scale (GES) | Immediately after / as soon as possible after the intervention (post-treatment)
  The General Self--Efficacy Scale (GES) is a self-report questionnaire used to measure self-efficacy. It is given to all study participants regardless of diagnosis. Total score values range from 10 to 40, with higher scores indicating a better outcome.
General Self--Efficacy Scale (GES) | 1-month follow-up
  The General Self--Efficacy Scale (GES) is a self-report questionnaire used to measure self-efficacy. It is given to all study participants regardless of diagnosis. Total score values range from 10 to 40, with higher scores indicating a better outcome.
Internal, Powerful Others, and Chance Questionnaire (IPC) | Baseline (pre-treatment)
  The Internal, Powerful Others, and Chance Questionnaire (IPC) is a self-report questionnaire used to measure locus of control. It is given to all study participants regardless of diagnosis. Score values of each of the three subscales range from 8 to 48, with higher scores on the subscale of internal orientation indicating a better outcome and higher scores on the subscales of powerful others orientation and chance orientation indicating a worse outcome.
Internal, Powerful Others, and Chance Questionnaire (IPC) | During the intervention (mid-treatment)
  The Internal, Powerful Others, and Chance Questionnaire (IPC) is a self-report questionnaire used to measure locus of control. It is given to all study participants regardless of diagnosis. Score values of each of the three subscales range from 8 to 48, with higher scores on the subscale of internal orientation indicating a better outcome and higher scores on the subscales of powerful others orientation and chance orientation indicating a worse outcome.
Internal, Powerful Others, and Chance Questionnaire (IPC) | Immediately after / as soon as possible after the intervention (post-treatment)
  The Internal, Powerful Others, and Chance Questionnaire (IPC) is a self-report questionnaire used to measure locus of control. It is given to all study participants regardless of diagnosis. Score values of each of the three subscales range from 8 to 48, with higher scores on the subscale of internal orientation indicating a better outcome and higher scores on the subscales of powerful others orientation and chance orientation indicating a worse outcome.
Internal, Powerful Others, and Chance Questionnaire (IPC) | 1-month follow-up
  The Internal, Powerful Others, and Chance Questionnaire (IPC) is a self-report questionnaire used to measure locus of control. It is given to all study participants regardless of diagnosis. Score values of each of the three subscales range from 8 to 48, with higher scores on the subscale of internal orientation indicating a better outcome and higher scores on the subscales of powerful others orientation and chance orientation indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Pyrkosch, Dipl.-Psych., Principal Investigator — Department of Psychiatry and Psychotherapy, Charité Campus Mitte - Universitätsmedizin Berlin; Anna Wehrheim, M.Sc.-Psych., Principal Investigator — Department of Psychiatry and Psychotherapy, Charité Campus Mitte - Universitätsmedizin Berlin
Locations (1):
- Department of Psychiatry and Psychotherapy, Charité Campus Mitte - Universitätsmedizin Berlin, Berlin, Germany